CLINICAL TRIAL: NCT03771053
Title: Intravascular Ultrasound Evaluation of the Intervention Effect of Simvastatin Combined With Ezetimibe on Coronary Borderline Lesion in Patients With Stable Angina Pectoris and Diabetes Mellitus Compared With Simvastatin Alone
Brief Title: The Effect of Simvastatin Combined With Ezetimibe in Patients With Stable Angina and Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, associate chief physician, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017FC-TSYS-3042
Record Dates: First submitted 2018-12-04; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; Atherosclerosis; Acute myocardial infarction; Coronary intervention
MeSH Terms: conditions — Coronary Disease; Atherosclerosis | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ezetimibe with simvastatin group (Experimental): ezetimibe 10mg with simvastatin 40mg everyday for 12 months after PCI
  Interventions: Drug: Ezetimibe with simvastatin
- Simvastatin group (Active Comparator): simvastatin 40mg everyday for 12 months after PCI
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Ezetimibe with simvastatin — ezetimibe 10mg with simvastatin 40mg everyday for 12 months after PCI
  Arms: Ezetimibe with simvastatin group
Drug: Simvastatin — simvastatin 40mg everyday for 12 months after PCI
  Arms: Simvastatin group

SUMMARY:
In this study, simvastatin combined with Ezeimebum was used to enhance lipid reduction, and IVUS was used to evaluate the volume and composition of coronary plaque before and after treatment. The aim is to evaluate the overall intervention effect of Ezeimebum on stable angina pectoris with diabetes mellitus on the basis of statins.

DETAILED DESCRIPTION:
This study was conducted in patients with stable angina pectoris complicated with diabetes mellitus in Chinese PLA General Hospital and coronary arteriography confirmed as critical lesion of coronary artery. The patients were randomly divided into two groups: ezeimebum combined with simvastatin group and simvastatin group. The patients of the former group were given ezeimebum 10mg combined with simvastatin 40mg for 12 months while the patients of the latter group were given simvastatin 40mg for 12 months. Assessed coronary atherosclerotic plaque volume percentage (PAV) and standardized total atherosclerotic plaque volume (TAV) by intravascular ultrasound (IVUS) at the time of entry and out of the group after 12 months. The changes of PAV level in both groups were taken as the main endpoints, and the changes of TAV levels in the two groups as the secondary endpoints. The changes of serum lipids and hypersensitive C-reactive protein levels were compared between the two groups before and after the treatment. Major cardiovascular events (non-fatal myocardial infarction, all-cause death, readmission to acute heart failure, and revascularization of recurrent angina pectoris) were followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-75 years
* consistent with the Chinese criteria for the diagnosis of chronic stable angina pectoris, stable angina pectoris symptoms in the last three months, and no more than CCS grade 3 of angina pectoris
* coronary angiography showed that the degree of coronary artery stenosis was 50% and 70%
* LDL-C standard: LDL-C > 80 mg/dL (2.08 mmol/L)
* The patients diagnosed with type 2 diabetes were currently using hypoglycemic drugs or insulin
* Sign the informed consent to join the group.

Exclusion Criteria:

* Acute coronary syndromes such as myocardial infarction, unstable angina pectoris, variant angina pectoris, cardiac shock, chronic heart failure, malignant arrhythmia, etc.
* Patients requiring stent implantation had been treated with intensive statins prior to admission (e.g. doses of Atto vastatin 40mg or resuvastatin 20mg)
* There were contraindications or statins for statin lowering lipids or statins, and there was a history of adverse reactions (liver injury, rash, myolysis, etc.) in the use of Ezeimebum, etc.
* Severe liver and kidney dysfunction, creatinine clearance < 30ml / min, acute pancreatitis, malignant tumor, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline coronary plaque volume percentage(PAV) at 12 months | 12 months after PCI
  PAV=∑（(ESA CSA-lumen CSA)/(ESA CSA)）x100, EEM CSA：cross-sectional area of outer elastic membrane boundary; lumen CSA: cross-sectional area of tube boundary

SECONDARY OUTCOMES:
Change from Baseline standardized coronary plaque volume(TAV) at 12 months | 12 months after PCI
  TAV= (median number of images in ∑ (ESA CSA-lumen CSA) / retracement) x number of images (standardized according to the length of IVUS retracement, To ensure that each individual patient has the same weight)
LDL-C | follow up in one year
  Low density lipoprotein cholesterol (LDL-C)
HDL-C | follow up in one year
  High density lipoprotein cholesterol (HDL-C)
TG | follow up in one year
  Total triglyceride(TG)
TC | follow up in one year
  Total cholesterol (TC)
Inflammation marker | follow up in one year
  hs-CRP

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Zhang X, Khan AA, Haq EU, Rahim A, Hu D, Attia J, Oldmeadow C, Ma X, Ding R, Boyle AJ. Increasing mortality from ischaemic heart disease in China from 2004 to 2010: disproportionate rise in rural areas and elderly subjects. 438 million person-years follow-up. Eur Heart J Qual Care Clin Outcomes. 2017 Jan 1;3(1):47-52. doi: 10.1093/ehjqcco/qcw041. PMID 28927191
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] Califf RM, Harrington RA, Blazing MA. Premature release of data from clinical trials of ezetimibe. N Engl J Med. 2009 Aug 13;361(7):712-7. doi: 10.1056/NEJMsr0900910. No abstract available. PMID 19675335
- [Background] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Background] Stein E, Stender S, Mata P, Sager P, Ponsonnet D, Melani L, Lipka L, Suresh R, Maccubbin D, Veltri E; Ezetimibe Study Group. Achieving lipoprotein goals in patients at high risk with severe hypercholesterolemia: efficacy and safety of ezetimibe co-administered with atorvastatin. Am Heart J. 2004 Sep;148(3):447-55. doi: 10.1016/j.ahj.2004.03.052. PMID 15389231
- [Background] van der Graaf A, Cuffie-Jackson C, Vissers MN, Trip MD, Gagne C, Shi G, Veltri E, Avis HJ, Kastelein JJ. Efficacy and safety of coadministration of ezetimibe and simvastatin in adolescents with heterozygous familial hypercholesterolemia. J Am Coll Cardiol. 2008 Oct 21;52(17):1421-9. doi: 10.1016/j.jacc.2008.09.002. PMID 18940534
- [Background] Nicholls SJ, Sipahi I. Emerging role of intravascular ultrasound in the assessment of experimental anti-atherosclerotic therapies. Curr Med Chem. 2006;13(15):1727-34. doi: 10.2174/092986706777452498. PMID 16787216
- [Background] Nissen SE, Nicholls SJ, Sipahi I, Libby P, Raichlen JS, Ballantyne CM, Davignon J, Erbel R, Fruchart JC, Tardif JC, Schoenhagen P, Crowe T, Cain V, Wolski K, Goormastic M, Tuzcu EM; ASTEROID Investigators. Effect of very high-intensity statin therapy on regression of coronary atherosclerosis: the ASTEROID trial. JAMA. 2006 Apr 5;295(13):1556-65. doi: 10.1001/jama.295.13.jpc60002. Epub 2006 Mar 13. PMID 16533939
- [Background] Nicholls SJ, Borgman M, Nissen SE, Raichlen JS, Ballantyne C, Barter P, Chapman MJ, Erbel R, Libby P. Impact of statins on progression of atherosclerosis: rationale and design of SATURN (Study of Coronary Atheroma by InTravascular Ultrasound: effect of Rosuvastatin versus AtorvastatiN). Curr Med Res Opin. 2011 Jun;27(6):1119-29. doi: 10.1185/03007995.2011.570746. Epub 2011 Mar 30. PMID 21446892
- [Background] Nicholls SJ, Ballantyne CM, Barter PJ, Chapman MJ, Erbel RM, Libby P, Raichlen JS, Uno K, Borgman M, Wolski K, Nissen SE. Effect of two intensive statin regimens on progression of coronary disease. N Engl J Med. 2011 Dec 1;365(22):2078-87. doi: 10.1056/NEJMoa1110874. Epub 2011 Nov 15. PMID 22085316